CLINICAL TRIAL: NCT00191503
Title: Phase II Study of Gemcitabine and Pemetrexed in Primary Unknown Adenocarcinoma
Brief Title: Gemcitabine and Pemetrexed in Primary Unknown Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9508; H3E-CA-S070
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — Pemetrexed; Gemcitabine

INTERVENTIONS:
Drug: Pemetrexed
Drug: Gemcitabine

SUMMARY:
There is no standard treatment for the patient population being asked to participate in this study. Although one current regimen, used by some investigators, has a high rate of response compared to other therapies, it is associated with moderate to severe toxicity. As gemcitabine and pemetrexed have a broad range of activity against cancer it is reasonable to determine how active and safe they are against patients with this type of cancer.The objective of this study is to determine the anti-tumor activity of pemetrexed and gemcitabine in patients with this condition.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma
* No obvious primary on routine history, physical examination, and investigations
* Patients greater than or equal to 18 years of age
* ECOG Performance Status 0-1
* Patients requiring opioids for pain control must be on a fixed analgesic regimen aimed to provide adequate pain control with no more than 3 breakthrough (supplemental) doses of analgesics per day to control pain; Additional inclusion criteria due apply, but not are not listed here.

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Unable to stabilize pain and analgesics for a period of 7 days prior to starting study treatment
* Prior treatment with chemotherapy
* Bilirubin greater than or equal to 40 mol/L
* AST or ALT greater than or equal to 5 times the upper limit of normal (ULN); Additional exclusion criteria due apply, but not are not listed here.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-01; Study Completion 2005-11

PRIMARY OUTCOMES:
The primary purpose of this study is to determine the objective response rate (ORR) for pemetrexed and gemcitabine when administered every two weeks to patients with adenocarcinoma of unknown origin who present with predominant liver metastases.

SECONDARY OUTCOMES:
The secondary objectives include measures of disease control including overall survival and to describe the toxicities of therapy in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9am - 5pm Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Edmonton, Alberta